CLINICAL TRIAL: NCT04853303
Title: The Use of a Virtual Reality Device (HypnoVR®) to Improve Chemotherapy-induced Nausea and Vomiting, Sleep Quality and Pain Among Children With Cancer in Hong Kong
Brief Title: VR to Improve CINV, Sleep and Pain Among Children With Cancer in HK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hypnoVR-NVSP
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Neoplasms; Child; Nausea; Vomiting; Sleep Hygiene; Pain
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting; Sleep Hygiene; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis VR (Experimental): The experimental group will receive a 15-minute hypnosis using virtual reality when they are experiencing chemotherapy-induced nausea and vomiting, sleep quality or pain.
  Interventions: Device: Hypnosis VR
- Control (No Intervention): The control group will receive no intervention.

INTERVENTIONS:
Device: Hypnosis VR — Children will be required to wear a VR gadget for hypnosis when they are experiencing chemotherapy-induced nausea and vomiting, sleep quality or pain. The duration is 15 minutes.
  Arms: Hypnosis VR

SUMMARY:
Chemotherapy-induced nausea and vomiting, sleep quality and pain are the common symptoms experienced by children with cancer. These symptoms significantly devastate the children's quality of life. Hypnosis is found to be effective in managing chemotherapy-induced nausea and vomiting, sleep quality and pain in children with cancer. In addition, virtual reality is shown to promote the effectiveness of hypnosis in managing these symptoms. However, no study so far has examine it effectiveness in Hong Kong Chinese children with cancer. This study aims to investigate the effectiveness in the use a virtual reality device to improve chemotherapy-induced nausea and vomiting, sleep quality and pain among children with cancer in Hong Kong.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. We recruit 180 children with cancer who are aged 9 to 18 and Chinese speaking and allocate them into experimental and control group. The experimental group will receive a 15-minute hypnosis using virtual reality when they are experiencing chemotherapy-induced nausea and vomiting, sleep quality or pain. The control group will receive no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 18
* Can read Chinese and speak Cantonese
* diagnosed with cancer

Exclusion Criteria:

* with mental disabilities or cognitive dysfunction as identified in the medical record

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Pediatric Nausea Assessment Tool (PeNAT) at the 6-month follow-up | at the 6-month follow-up
  Children will be required o fill in the Chinese version of the Pediatric Nausea Assessment Tool (PeNAT) at 6-month follow-up. The score ranges from 1 to 4. Higher scores represent a more severe nausea.
Pittsburgh Sleep Quality Index (PSQI) at the 6-month follow-up | at the 6-month follow-up
  Children will be required to fill in the Pittsburgh Sleep Quality Index (PSQI) at the 6-month follow-up. The score ranges from 0 to 21. Higher scores represent to poorer sleep quality.
Visual Analogue Pain Scale (VAS) at the 6-month follow-up | at the 6-month follow-up
  Children will be required to fill in the Visual Analogue Pain Scale (VAS) at 6-month follow-up. The score ranges from 0 to 10. Higher scores represent a higher level of pain.

SECONDARY OUTCOMES:
The Pediatric Nausea Assessment Tool (PeNAT) at baseline | at baseline
  Children will be required to fill in the Chinese version of the Pediatric Nausea Assessment Tool (PeNAT) at baseline. The score ranges from 1 to 4. Higher scores represent a more severe nausea.
The Pediatric Nausea Assessment Tool (PeNAT) at 1-month follow-up | at 1-month follow-up
  Children will be required to fill in the Chinese version of the Pediatric Nausea Assessment Tool (PeNAT) at 1-month follow-up.The score ranges from 1 to 4. Higher scores represent a more severe nausea.
The Pediatric Nausea Assessment Tool (PeNAT) at 3-month follow-up | at 3-month follow-up
  Children will be required to fill in the Chinese version of the Pediatric Nausea Assessment Tool (PeNAT) at 3-month follow-up. The score ranges from 1 to 4. Higher scores represent a more severe nausea.
Pittsburgh Sleep Quality Index (PSQI) at baseline | at baseline
  Children will be required to fill in the Pittsburgh Sleep Quality Index (PSQI) at baseline. The score ranges from 0 to 21. Higher scores represent to poorer sleep quality.
Pittsburgh Sleep Quality Index (PSQI) at 1-month follow-up | at 1-month follow-up
  Children will be required to fill in the Pittsburgh Sleep Quality Index (PSQI) at 1-month follow-up. The score ranges from 0 to 21. Higher scores represent to poorer sleep quality.
Pittsburgh Sleep Quality Index (PSQI) at 3-month follow-up | at 3-month follow-up
  Children will be required to fill in the Pittsburgh Sleep Quality Index (PSQI) at 3-month follow-up. The score ranges from 0 to 21. Higher scores represent to poorer sleep quality.
Visual Analogue Pain Scale (VAS) at baseline | at baseline
  Children will be required to fill in the Visual Analogue Pain Scale (VAS) at baseline. The score ranges from 0 to 10. Higher scores represent a higher level of pain.
Visual Analogue Pain Scale (VAS) at 1-month follow-up | at 1-month follow-up
  Children will be required to fill in the Visual Analogue Pain Scale (VAS) at 1-month follow-up. The score ranges from 0 to 10. Higher scores represent a higher level of pain.
Visual Analogue Pain Scale (VAS) at 3-month follow-up | at 3-month follow-up
  Children will be required to fill in the Visual Analogue Pain Scale (VAS) at 3-month follow-up. The score ranges from 0 to 10. Higher scores represent a higher level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No